CLINICAL TRIAL: NCT00427206
Title: Hepatic Function Following Five Days of Therapeutic Dosing of Acetaminophen in Alcoholics
Brief Title: Hepatic Function in Alcoholics Following 5 Days of Acetaminophen Dosing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: COMIRB #04-0486
Record Dates: First submitted 2007-01-24; First posted 2007-01-26 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-02

CONDITIONS: Alcohol Related Disorders
Keywords: acetaminophen; alcohol; liver injury
MeSH Terms: conditions — Alcohol-Related Disorders | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): acetaminophen 4 g/day
  Interventions: Drug: acetaminophen (4g/day)
- 2 (Placebo Comparator): placebo undistinguishable from active drug
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: acetaminophen (4g/day)
  Arms: 1
Drug: placebo
  Arms: 2

SUMMARY:
The study objective was to determine if liver injury develops in alcoholic patients during or following 5 days of therapeutic acetaminophen dosing. Volunteers were recruited from two community detoxification centers to take either acetaminophen (4g/day) or placebo for 5 consecutive days. All subjects were monitored an additional two days following the dosing period. The primary measures were aminotransferase measures taken at baseline and Days 2, 4, 6 and 7. We hypothesized that there would be no difference in aminotransferase means between the groups at any study period.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* admitted to participating detox facility with a positive BAL at the time of admittance
* signed a written informed consent

Exclusion Criteria:

* serum acetaminophen level greater than 20 mcg/ml
* serum AST or ALT levels greater than 200 IU/L
* INR greater than 1.5
* if female, positive for beta-subunit of chorionic gonadotropin (beta-HCG)
* clinically intoxicated, psychiatrically impaired or unable to give informed consent
* known hypersensitivity to acetaminophen
* history of ingesting more than four grams of APAP per day for any of the four days preceding study enrollment
* currently enrolled in another trial or had been enrolled in another trial in the preceding three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2004-11; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
group mean aminotransferase measures
mean change in aminotransferase measures between study groups

SECONDARY OUTCOMES:
proportion of subjects that develop an aminotransferase level greater than the upper limit of reference range
proportion of subjects that develop hepatotoxicity (ALT>1000 IU/L)
proportion of subjects that develop drug induced liver injury

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Dart, MD, PhD, Principal Investigator — Denver Health/Rocky Mountain Poison & Drug Center; Bruna Brands, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (2):
- Denver CARES, Denver, Colorado, United States
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada